CLINICAL TRIAL: NCT04473508
Title: Erectus Nerve Block for Lumbar Spine Surgery : a Prospective Randomized Study
Brief Title: Erectus Nerve Block for Lumbar Spine Surgery
Acronym: EFABE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOCAL/2018/PC-02; 2019-001678-26 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-07-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-03

CONDITIONS: Spine Surgery; Pain Relief; Morphine; AdverseEvent
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Experimental): active treatment (Local anaesthetic): Local administration of ropivacaine 30 mL (5mg/mL)
  Interventions: Drug: Local administration of ropivacaine
- Control (Placebo Comparator): Local administration of Placebo ( Saline Solution)
  Interventions: Drug: Local administration of placebo (saline solution)

INTERVENTIONS:
Drug: Local administration of ropivacaine — Erector nerve block with local ropivacaine injection in addition with conventional anesthesia for spine surgery
  Arms: Treated
Drug: Local administration of placebo (saline solution) — injection of saline solution in addition with conventional anesthesia for spine surgery
  Arms: Control

SUMMARY:
: Spine surgery induced severe postoperative pain. Several techniques as intravenous multimodal analgesia have been proposed to reduce pain relief and morphine rescue over the first postoperative days. Regional anesthesia using the erectus nerve block is a simple infiltration across lamina of the vertebra: Ultrasound-guided posterior ramus of spinal nerve block for anesthesia and analgesia in lumbar spinal surgery This study compared erector nerve block with local anesthetic vs placebo to reduce pain and morphine rescue after lumbar spine surgery. The investigators hypothesized that eructor nerve block induced a large block from L1 to L5 that induced posterior nerve roots block anesthesia. This block reduced pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age> 18years and <80 years
* lumbar spine surgery (2-4 levels)
* posterior approach
* ASA 1-3

Exclusion Criteria:

* refusal
* age < 18yrs
* <50 kg and >120 kg
* pregnant
* renal or hepatic severe desease
* ASA 4
* no French speaking
* emergency surgery
* local or systemic infection
* surgical resumption of the surgical site
* surgery involving a thoracic approach
* allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
morphine consumption (mg) | 24 Hours after surgery
  Quantity administered in the post-interventional monitoring room and in hospitalization via a self-controlled morphine pump by the patient

SECONDARY OUTCOMES:
Adverse events | from surgery to 3 months
  Nausea, vomiting, confusion, urinary retention, hematoma, reintervention
pain at rest and at movement: Visual Analogic scale | Day 1 to Day 3, Day od hospital discharge and month 3
  Visual Analogic scale of pain (0-10)
chronic pain: DN4 questionnaire | Questionnaire DN4 at 3 months
  pain score as mesured with DN4 questionnaire
Length of hospital stay | hospital length of stay, an average of 4 days
  Number of day in hospital
Length of stay in the post-intervention care unit | Day 1
  Number of minutes that patient stay in post intervention care unit in minutes
Patient Satisfaction: visual analogic scale | Day of hospital discharge, an average of day 4
  Patient satisfaction mesured with a visual analogic scale (0-10)
Patient Quality of life: EQ-5D Questionnaire | 3 months
  Patient Quality of life mesured with EQ-5D Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Avis, Md, Principal Investigator — Geoffrey.avis@chu-nimes.fr
Locations (1):
- CHU Nimes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avis G, Gricourt Y, Vialatte PB, Meunier V, Perin M, Simon N, Claret PG, El Fertit H, Lefrant JY, Bertrand M, Cuvillon P. Analgesic efficacy of erector spinae plane blocks for lumbar spine surgery: a randomized double-blind controlled clinical trial. Reg Anesth Pain Med. 2022 Jul 21:rapm-2022-103737. doi: 10.1136/rapm-2022-103737. Online ahead of print. PMID 35863786